CLINICAL TRIAL: NCT02119572
Title: Impact of Peer Support on Diabetes in China: a Multi-center, Cluster Randomized Controlled Trial
Brief Title: Impact of Peer Support on Diabetes in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, director of endocrine department, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: Zhongdaendo1
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes
Keywords: diabetes,peer support
MeSH Terms: conditions — Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peer support (Experimental): Patients are divided into small groups and assigned with peer leaders for twelve months according to their residence. Besides the same training and follow-ups as the control arm, patients from intervention groups are suggested and encouraged to take part in the group activities with the peer leaders per month. And if possible, casual activities (such as phone call, chatting, short message; physical exercise, group member family visiting，going to supermarket together, etc.)are also recommended
  Interventions: Behavioral: peer support; Other: usual education lectures
- usual education (Active Comparator): Patients attend the usual self-management education and communicate with the professionals every two months, getting the information on diabetes diet, exercise, glucose monitor, etc. besides that the group members should attend three follow ups at baseline,6 and 12 months.
  Interventions: Other: usual education lectures

INTERVENTIONS:
Behavioral: peer support
  Other Names: peer education, peer coach
  Arms: peer support
Other: usual education lectures

SUMMARY:
The prevalence of diabetes has been growing rapidly in developing countries causing a devastating economic burden and increasing demands on healthcare systems. Therefore, there is an urgent need to find cost-effective and multi-faceted approach for diabetes care. Peer support models provide a potentially low-cost, flexible means that is complimentary to the current existing health care services. Trained peer leaders can become qualified extenders to a formal healthcare system, thereby, assisting with the education delivery and bolstering the efforts of the professional staff. To implement a culturally- specific peer support program and determine whether it is acceptable, cost-effective in China is important. This study aims to implement and evaluate biophysical and psychosocial outcomes of a peer support program and to explore it's feasibility and sustainability in China

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. with voluntary participation and have signed the Patient Informed Consent Sheet
3. reside in stable places during the intervention period

Exclusion Criteria:

1. Patients with reduced life expectancy and unstable mood or major psychiatric conditions
2. suffering from cancer and have been receiving radiotherapy and/ or chemotherapy in the past half year
3. enrolling in other research program at present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 6 months,12 months | baselline,6months,12months

SECONDARY OUTCOMES:
Change from Baseline blood pressure at 6 months,12 months | baseline,6 months,12months
Change from Baseline months BMI at 6 months,12 months | baseline,6 months,12months
Change from Baseline months blood liquids at 6 months,12 months | baseline,6 months,12months
Change from Baseline months blood glucose at 6 months,12 months | baseline,6 months,12months
Change from baseline in diabetes self-care activities scales at 6 months,12months | baseline,6 months,12months
Change from baseline in depression scales at 6 months,12months | baseline,6 months,12months
Change from baseline in medication adherence scales at 6 months,12months | baseline,6 months,12months
Change from baseline in quality of life scales at 6 months,12months | baseline,6 months,12months
Change from baseline in diabetes self-efficacy scales at 6 months,12months | baseline,6 months,12months
Change from baseline in diabetes knowledge scales at 6 months,12months | baseline,6 months, 12 months
Change from baseline in positive and negative affectivity at 6 months,12months | baseline, 6 months,12months
Change from baseline in events of hypoglycemia at 6 months,12months | baseline,6 months,12months
Change from baseline advanced glycation end products at 6 months,12months | baseline ,6 months,12months
cost | baseline,6 months,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zilin Sun, Dr., Principal Investigator — Zhongda Hospital
Locations (1):
- Liuhe, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ju C, Shi R, Yao L, Ye X, Jia M, Han J, Yang T, Lu Q, Jin H, Cai X, Yuan S, Xie B, Yu X, Coufal MM, Fisher EB, Sun Z. Effect of peer support on diabetes distress: a cluster randomized controlled trial. Diabet Med. 2018 Jun;35(6):770-775. doi: 10.1111/dme.13625. Epub 2018 Apr 11. PMID 29574995
- [Derived] Xie B, Ye XL, Sun ZL, Jia M, Jin H, Ju CP, Yao L, De Vladmir CH, Yang Y. Peer support for patients with type 2 diabetes in rural communities of China: protocol for a cluster randomized controlled trial. BMC Public Health. 2014 Jul 23;14:747. doi: 10.1186/1471-2458-14-747. PMID 25056813